CLINICAL TRIAL: NCT00566839
Title: Randomized Comparison of Thoracoscopic Lung Volume Reduction Surgery Performed by Resectional Surgical Technique Under General Anesthesia or by a Non-Resectional Technique in Awake Patients Under Sole Epidural Anesthesia
Brief Title: Randomized Comparison of Awake Nonresectional Versus Nonawake Resectional Lung Volume Reduction Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Tommaso Claudio Mineo, Tor Vergata University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MED2112025; enfis12022
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Last update posted 2007-12-04 (Estimated); Status verified 2007-10

CONDITIONS: Pulmonary Emphysema
Keywords: COPD; LVRS; Awake surgery; Thoracic epidural anesthesia; One-lung ventilation; Emphysema; VATS; Lung surgery
MeSH Terms: conditions — Pulmonary Emphysema; Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: awake nonresectional LVRS
- 2 (Active Comparator)
  Interventions: Procedure: Nonawake resectional LVRS

INTERVENTIONS:
Procedure: awake nonresectional LVRS — Thoracoscopic nonresectional lung volume reduction surgery carried out in awake patients under sole epidural anesthesia through plication of most emphysematous target areas of the lung
  Arms: 1
Procedure: Nonawake resectional LVRS — Thoracoscopic lung volume reduction surgery carried out under general anesthesia and one-lung ventilation through nonanatomic resection of the most emphysematous target areas of the lung
  Arms: 2

SUMMARY:
Lung volume reduction surgery is effective in improving pulmonary function and quality of life in selected patients with severe emphysema although the morbidity of this surgical procedure is still considerable. Morbidity is mainly addressed to general anesthesia-related adverse effects and surgical trauma deriving from lung resection. Having developed an awake nonresectional lung volume reduction surgery technique, which is performed under sole thoracic epidural anesthesia, we have hypothesized that it could offer satisfactory clinical results and reduced morbidity rate when compared with the conventional surgical procedure.

DETAILED DESCRIPTION:
There is increasing scientific evidence that resectional lung volume reduction (LVR) can induce long lasting clinical improvements in selected patients with upper-lobe predominant emphysema and that clinical benefit and survival are better than those achieved with maximized medical treatment. The most widely employed surgical technique entails unilateral or bilateral staple resection of the most emphysematous lung tissue performed under general anesthesia through open or thoracoscopic approaches.

However, the type of surgical approach did not modify the considerable procedure-related morbidity, which can be mainly addressed to general anesthesia and surgical trauma deriving from resection of emphysematous lung tissue. Indeed, following resectional LVR expected mortality and pulmonary morbidity are 5.5% and 30%, respectively. Time spent for postoperative recovering is often prolonged with about 30% of patients still hospitalized or in rehabilitation facilities at 1 month and 15% still not at home 2 months after the operation. As a result, the cost-effectiveness of LVR continue to be questioned.

In recent years, the concept of nonresectional LVR is being investigated and new bronchoscopic approaches have been developed in an attempt of reducing the typical shortcomings of resectional LVR. Within the framework of the proposed nonsurgical methods which differ somewhat in physiopathologic bases and mechanism of LVR, a common denominator is that, so far, all needed general anesthesia.

We have developed an awake nonresectional LVR surgery technique, which respects the basic concepts of resectional LVR but adds some theoretical advantages and is performed under sole thoracic epidural anesthesia.

Following an initial pilot study to assess feasibility and early results, we want to analyze in a randomized fashion the perioperative morbidity and comprehensive 2-year results of thoracoscopic lung volume reduction surgery performed by the awake nonresectional or nonawake resectional surgical techniques.

ELIGIBILITY:
Inclusion Criteria:

* Severe smoking-related emphysema with upper-lobe predominance
* Severe disability (MMRC dyspnea grade>=3) despite maximized medical therapy including respiratory rehabilitation
* No clinically significant sputum production, bronchiectasis or asthma postbronchodilator forced expiratory volume in onee second (FEV1)<40% predicted
* Residual volume (RV)>180% predicted at body plethysmography
* Total Lung capacity>120% predicted
* No instable angina or ventricular arrythmia
* Peak systolic pulmonary artery pressure <50 mmHg at echocardiocolordoppler
* Arterial carbon dioxide (PaCO2)<50 mmHg
* Diffusion capacity of carbon monoxide (DLCO)> 20% predicted
* Quit smoking since at least 4 months
* ASA score<=3
* Body mass index >18 <29
* No comorbid condition that would significantly increase operative risk or negatively affect participation in a vigorous respiratory rehabilitation program
* No neoplastic disease with life expectancy < 12 months
* No previous pleurodesis or thoracotomy in the more affected hemithorax

Exclusion Criteria:

* Radiologic evidence of extensive pleural adhesions with pleural scarring and calcifications on site targeted for LVRS
* Patients refusal or noncompliance to thoracic epidural anesthesia and awake surgery
* Patients refusal or noncompliance to general surgery and one-lung ventilation
* Unfavorable anatomy for thoracic epidural anesthesia
* Previous surgery of the cervical or upper thoracic spine
* Compromised coagulation (thromboplastin time<80%, prothrombin time>40 sec, platelet count<100/nL or bleeding disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-12; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
mortality | 3 months
Hospital stay | 2 months
Forced expiratory volume in one second | 24 months
Residual volume | 24 months
Modified Medical research Council Dyspnea index | 24 months

SECONDARY OUTCOMES:
Arterial carbon dioxide tension (mmHg) | 2 days
Arterial oxygen to fraction of inspired oxygen ratio (PaO2/FiO2) | 2 days
Anesthesia satisfaction score (graded from 1=unsatisfactory to 4=Excellent) | 1 day (24h post-surgery)
Six minute walking test distance (m) | 24 months
Short form 36-item quality of life physical function domain score | 24 months
Body mass index (Kg/m2) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Pompeo, MD, Principal Investigator — Thoracic Surgery Division, Policlinico Tor Vergata University; Tommaso C Mineo, MD, Study Chair — Thoracic Surgery Division, Policlinico Tor Vergata University
Locations (1):
- Policlinico Tor Vergata University, Rome, Italy

REFERENCES:
- [Background] Pompeo E, Marino M, Nofroni I, Matteucci G, Mineo TC. Reduction pneumoplasty versus respiratory rehabilitation in severe emphysema: a randomized study. Pulmonary Emphysema Research Group. Ann Thorac Surg. 2000 Sep;70(3):948-53; discussion 954. doi: 10.1016/s0003-4975(00)01646-5. PMID 11016339
- [Background] Mineo TC, Pompeo E, Rogliani P, Dauri M, Turani F, Bollero P, Magliocchetti N. Effect of lung volume reduction surgery for severe emphysema on right ventricular function. Am J Respir Crit Care Med. 2002 Feb 15;165(4):489-94. doi: 10.1164/ajrccm.165.4.2108129. PMID 11850341
- [Background] Pompeo E, Mineo TC; Pulmonary Emphysema Research group. Long-term outcome of staged versus one-stage bilateral thoracoscopic reduction pneumoplasty. Eur J Cardiothorac Surg. 2002 Apr;21(4):627-33; discussion 633. doi: 10.1016/s1010-7940(02)00038-6. PMID 11932158
- [Background] Mineo TC, Ambrogi V, Pompeo E, Bollero P, Mineo D, Nofroni I; Pulmonary Emphysema Research Group. Body weight and nutritional changes after reduction pneumoplasty for severe emphysema: a randomized study. J Thorac Cardiovasc Surg. 2002 Oct;124(4):660-7. doi: 10.1067/mtc.2002.123807. PMID 12324722
- [Background] Pompeo E, De Dominicis E, Ambrogi V, Mineo D, Elia S, Mineo TC. Quality of life after tailored combined surgery for stage I non-small-cell lung cancer and severe emphysema. Ann Thorac Surg. 2003 Dec;76(6):1821-7. doi: 10.1016/s0003-4975(03)01302-x. PMID 14667591
- [Background] Mineo TC, Ambrogi V, Pompeo E, Elia S, Mineo D, Bollero P, Nofroni I. Impact of lung volume reduction surgery versus rehabilitation on quality of life. Eur Respir J. 2004 Feb;23(2):275-80. doi: 10.1183/09031936.03.00025203. PMID 14979503
- [Background] Mineo TC, Pompeo E, Mineo D, Rogliani P, Leonardis C, Nofroni I. Results of unilateral lung volume reduction surgery in patients with distinct heterogeneity of emphysema between lungs. J Thorac Cardiovasc Surg. 2005 Jan;129(1):73-9. doi: 10.1016/j.jtcvs.2004.05.024. PMID 15632827
- [Background] Tacconi F, Pompeo E, Mineo TC. Late-onset occult pneumothorax after lung volume-reduction surgery. Ann Thorac Surg. 2005 Dec;80(6):2008-12. doi: 10.1016/j.athoracsur.2005.06.013. PMID 16305835
- [Background] Mineo TC, Pompeo E, Mineo D, Tacconi F, Marino M, Sabato AF. Awake nonresectional lung volume reduction surgery. Ann Surg. 2006 Jan;243(1):131-6. doi: 10.1097/01.sla.0000182917.39534.2c. PMID 16371748
- [Background] Mineo TC, Pompeo E, Mineo D, Ambrogi V, Ciarapica D, Polito A. Resting energy expenditure and metabolic changes after lung volume reduction surgery for emphysema. Ann Thorac Surg. 2006 Oct;82(4):1205-11. doi: 10.1016/j.athoracsur.2006.05.030. PMID 16996909
- [Background] Mineo TC, Pompeo E. Long-term results of tailored lung volume reduction surgery for severe emphysema. Clin Ter. 2007 Mar-Apr;158(2):127-33. PMID 17566513
- [Background] Pompeo E, Mineo TC. Two-year improvement in multidimensional body mass index, airflow obstruction, dyspnea, and exercise capacity index after nonresectional lung volume reduction surgery in awake patients. Ann Thorac Surg. 2007 Dec;84(6):1862-9; discussion 1862-9. doi: 10.1016/j.athoracsur.2007.07.007. PMID 18036900
- [Derived] Pompeo E, Rogliani P, Tacconi F, Dauri M, Saltini C, Novelli G, Mineo TC; Awake Thoracic Surgery Research Group. Randomized comparison of awake nonresectional versus nonawake resectional lung volume reduction surgery. J Thorac Cardiovasc Surg. 2012 Jan;143(1):47-54, 54.e1. doi: 10.1016/j.jtcvs.2011.09.050. Epub 2011 Nov 4. PMID 22056369